CLINICAL TRIAL: NCT06810206
Title: A Comparison Between The Efficacy of Modified Thoracoabdominal Plane Block Via Perichondral Approach (M-TAPA) And External Oblique Intercostal Plane Block (EOIPB) in Patients Undergoing Laparoscopic Cholecystectomy Surgeries (LC): A Double-Blinded Randomized Comparative Study.
Brief Title: A Comparison Between The Efficacy of Modified Thoracoabdominal Plane Block Via Perichondral Approach (M-TAPA) And External Oblique Intercostal Plane Block (EOIPB) in Patients Undergoing Laparoscopic Cholecystectomy Surgeries (LC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Miran Mohamed Abdelmagyd, Doctor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD-462-2024
Record Dates: First submitted 2025-01-26; First posted 2025-02-05 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Post Operative Pain
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, randomized comparative study with two parallel groups. Participants will be randomly assigned to receive either the MTAPA or the EOIPB.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: 30 patients will receive the MTAPA.
  Interventions: Other: Bilateral Ultrasound Guidance M-TAPA
- Group B (Active Comparator): Group B: 30 patients will receive the EOIPB.
  Interventions: Procedure: Bilateral Ultrasound Guidance EOIPB

INTERVENTIONS:
Other: Bilateral Ultrasound Guidance M-TAPA — transversus abdominis, internal oblique, and external oblique muscles will be identified on the costochondral angle in the sagittal plane at the 10th costal margin. deep angle will be given to the costochondral angle at the edge of the 10th costa with the probe in the sagittal direction to view the lower surface of the costal cartilage in the midline. The needle will be inserted in the cranial direction using the in-plane technique, and the needle tip will be moved to the posterior aspect of the 10th costal cartilage, and saline (5 ml) will be injected to confirm the location by observing dissection between internal oblique muscle and transversus abdominis muscle under the 10th costal cartilage, and local anesthetic will be injected into the lower surface of the chondrium. The local anesthetic to be used is bupivacaine 0.25% with Ultrasound Siemens® ACUSON X300 portable scanner with a high frequency linear transducer (10 MHz) using A Quincke 22 G . x 3½ in. (0.7x88 mm) A spinal needle
  Other Names: Modified throacoabdominal plane block (M-TAPA); GROUP A
  Arms: Group A
Procedure: Bilateral Ultrasound Guidance EOIPB — The patients will be positioned in the supine position with the ipsilateral arm in abduction. The transducer will be positioned in a cephalad to caudad parasagittal plane at the anterior axillary line at the level of the sixth and seventh ribs in line with the xiphoid process. Using the in-plane technique, the needle will be advanced from cephalad to caudad until the tip lies in the plane between the external oblique muscle and intercostal muscles between the sixth and seventh ribs. Following hydro-dissection with 2 ml of 0.9% saline to confirm the correct needle tip position, LA injection will be given. The same procedure will then be repeated on the contralateral
  * Local anesthetics to be injected: iBupivacaine (0.25%)
  * Dose : 25ml on each side
  * Device to be used: Ultrasound Siemens® ACUSON X300 portable scanner with a high-frequency linear transducer (10 MHz) that is covered in sterile plastic.
  * Needle to be used : A Quincke 22 G . x 3½ inch (0.7x88 mm) spinal needle
  Other Names: External Oblique Intercoastal Plane Block ( EOIPB ); GROUP B
  Arms: Group B

SUMMARY:
Because laparoscopic procedures have a number of benefits over open procedures, they have completely changed the surgical industry.(1) Laparoscopic cholecystectomy (LC) is a minimally invasive technique that usually yields less discomfort following surgery, shorter hospital stays, and quicker patient recovery, plus it's an economical operation. Nevertheless, it results in moderate to severe pain.(2).By using regional anesthesia techniques to effectively control pain and lessen the requirement for opioid analgesics, ERAS implementation has demonstrated significant decreases in opioid usage and improved overall patient outcomes (3). (4) To minimize the need for opioids, opioid sparing anesthesia employs a multimodal strategy that includes nonsteroidal anti-inflammatory medications, paracetamol, local anesthetics (LA), and, if feasible, regional anesthetic techniques and regional analgesia. (5) With fewer systemic side effects, regional anesthetic techniques-like nerve blocks-offer tailored pain treatment. The best regional pain management strategy for LC surgery is still unknown, though.(4) Modified Thoracoabdominal Nerves Block Through Perichondral Approach (M-TAPA) Block is a new technique defined as a modification of TAPA Block in which local anaesthetics are administered only to the underside of the perichondral surface, creating a sensory block between T5-T12 dermatomes. While the external oblique intercostal plane (EOIPB) block provides blockade of the lateral and anterior cutaneous branches of the intercostal nerves from T6/7 to T10/11.This study aims to compare the efficacy of both MTAPA and EOIPB in patients undergoing LC surgery .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Scheduled for Laparoscopic cholecystectomy surgery
* ASA (American Society of Anaesthesiologists) physical status I-II

Exclusion Criteria:

* Known allergy to local anaesthetics
* Coagulopathy or anticoagulant use
* Infection at the site of block
* Chronic pain conditions
* Advanced liver or kidney failure
* History of abdominal surgery or trauma
* Alcohol or drug use
* Refusal to participate
* Chronic opioid consumption
* Use of painkillers in the preoperative 24hours
* Conversion to open surgery
* Body mass index ( BMI ) > 35

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
comparing the effectiveness of the modified thoracoabdominal plane block via perichondral approach versus the external oblique intercoastal plane block in reducing pain in laparoscopic cholecystectomy surgery's patients through calculating the mean NRS | . NRS scores will be recorded postoperatively upon arrival to PACU and it will be noted as point (0) and then at 20 minutes , and then after the 1st hour , and the at the 6th hour , 12 th hour and 24th hour for a total of 24-hour period.
  Numerical Rating Score (NRS) for Pain severity will be measured with a NRS of 0, being no pain , while of 10 being worst pain imaginable. NRS scores will be recorded postoperatively upon arrival to PACU and it will be noted as point (0) and then at 20 minutes , and then after the 1st hour , and the at the 6th hour , 12 th hour and 24th hour for a total of 24-hour period. (11) Patients will be educated and familiarized with NRS scores in the preoperative period. Postoperative, pain control regimen will be used for the two groups as Paracetamol 15mg/kg IV /6hours, Ketorolac 30mg IV /8hours. If the patient's NRS pain score happens to be ≥ 4 points, 10 mg of intravenous nalbuphine Will be given , and the NRS will be repeated again after 15 minutes , if still > 4 , additional 10 mg IV nalbuphine will be given , with maximum dose of 20 mg per dose , can be repeated up to four times per day with maximum dose of 80 mg per day (18)

SECONDARY OUTCOMES:
evaluating the quality of recovery via the QOR-40 questionnaire. | the Quality of Recovery-40 (QoR-40) questionnaire will be used in PACU after 10 minutes from patient arrival to the PACU .
  To evaluate the quality of recovery, the Quality of Recovery-40 (QoR-40) questionnaire will be used in PACU after 10 minutes from patient arrival to the PACU. Scores range from a minimum of 40 (poor recovery) to a maximum of 200 (excellent recovery).
identifying dermatomal coverage of each block via pinprick test. | Dermatomal coverage will be tested using pinprick test in PACU after evaluating the QoR-40 within the first hour postoperatively
  Dermatomal coverage will be tested using pinprick test to evaluate the T3-L1 sensory levels in PACU after evaluating the QoR-40 ( since block will be administered after induction of anaesthesia ) . Anterior and lateral cutaneous branches will be evaluated on a vertical line 3-5 cm from the midline and midaxillary lines, respectively. A 3-point numerical scale (0 = no pain, 1 = decreasing pain, 2 = normal pain) will be used. The values of 0 or 1 will be defined as effective . The normal sense in the shoulder will be used for comparison. (11,17)
evaluating the efficacy of each block in providing analgesia intraoperatively by measuring amount of fentanyl consumed in micrograms | intraoperatively
  * Anaesthesia induction and endotracheal intubation will be performed after preoxygenation with 100% oxygen, intravenously using propofol 2 mg/kg, fentanyl 1-2 µg/kg, and atracurium 0.5 mg/kg. Anaesthesia will be maintained with isoflurane (0.8-1.2 MAC) and atracurium 0.1mg/kg/20 mins
  * additional boluses of fentanyl IV dose of 0.25 micrograms/kg/dose will be given if blood pressure and/or heart rate increase by 20% of baseline, with calculation of total fentanyl consumption intraoperatively in micrograms
Total opioid consumption in the first 24 hours postoperatively in mgs | postoperatively with a total of 24 hour
  * Total Nalbuphine consumption will be recorded in mgs for a total of 24-hour period
  * Postoperative pain control regimen will be used for the two groups as Paracetamol 15mg/kg IV / 6 hours, Ketorolac 30 mg IV/8 hours. If the patient's NRS pain score happens to be ≥ 4 points, 10 mg of intravenous nalbuphine Will be given , and the NRS will be repeated again after 15 minutes , if still > 4; additional 10 mg IV nalbuphine will be given , with maximum dose of 20 mg per dose that can be repeated up to four times per day with maximum dose of 80 mg per day
Time to first mobilization in hours | postoperatively up to 24 hour
  ●The time to mobilization of the patients following surgery will be recorded in hours Mobilization will be defined as being able to at least sit on the edge of the bed.
Incidence of block-related complications | postoperatively with a total of 24 hour
  Incidence of block-related complications (e.g., hematoma, infection, nerve damage , LAST )
Incidence of PONV. | every six hours for a total of 24 hour postoperatively
  ●Verbal descriptive scale for Postoperative Nausea and Vomiting (PONV) will be used with 0 = none , 1 = mild nausea , 2= moderate nausea , 3= vomiting once , 4= multiple vomiting .
the Time to first rescue opioid | it will be measured postoperatively for a total period of 24 hour
  the time to first rescue opioid will be noted and defined as the duration in hours that the patient lasted without the need of nalbuphine IV dose of 10 mg (NRS<4).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of medicine , Kasr Al Aini Hospitals , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bilge A, Basaran B, Et T, Korkusuz M, Yarimoglu R, Toprak H, Kumru N. Ultrasound-guided bilateral modified-thoracoabdominal nerve block through a perichondrial approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy: a randomized double-blind controlled trial. BMC Anesthesiol. 2022 Oct 28;22(1):329. doi: 10.1186/s12871-022-01866-4. PMID 36307755